CLINICAL TRIAL: NCT05387603
Title: Systemic Targeted Adaptive RadioTherapy of NeuroEndocrine Tumors. An Open-label, Multicenter, Randomized Phase III Trial Comparing Safety and Efficacy of Personalized Versus Non-personalized Radionuclide Therapy With 177Lu (Lutetium)-DOTATOC.
Brief Title: Systemic Targeted Adaptive RadioTherapy of NeuroEndocrine Tumors.
Acronym: START-NET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: START-01; 2021-002218-15 (EudraCT Number)
Record Dates: First submitted 2022-04-21; First posted 2022-05-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine tumors; Radionuclide therapy; Personalized radionuclide therapy; 177Lu-DOTATOC; Capecitabine; Dosimetry-based radionuclide therapy; Somatostatin receptor; Lutetium; Beta- and gamma-emitting radionuclide; Translational research
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-; Capecitabine

STUDY DESIGN:
Intervention Model Description: This is a randomized, open-label, controlled trial in which patients are assigned to either non-personalized treatment with 4 cycles of 7.5 gigabequerel (GBq) 177Lu-DOTATOC (TOC), or personalized treatment based on dual imaging. In the personalized arm patients are treated according to the results of the dual imaging at screening:
  A. Patients with 68Ga-1,4,7,10-tetra-azacyclododecane-N.n,N,N-tetraacetic acid (DOTA)-positron emission tomography (PET)-positive but 18F-2-fluoro-2-deoxy-D-glucosefluorodeoxyglucose (FDG)-PET-negative NET will receive dosimetry-based PRRT only (dTOC) B. Patients with 68Ga-DOTA- and 18F-FDG-PET-positive NET will receive a combination of capecitabine and dosimetry-based PRRT (CAP-dTOC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 177Lu-DOTATOC + Capecitabine (Experimental): Patients with 68Ga-DOTA- and 18F-FDG-PET-positive NET will receive a combination of intravenous 7.5 GBG (gigabequerel) 177Lu-DOTATOC for about 7 cycles in combination with capecitabine (4 cycles, cycle length 3 weeks, with one week without capecitabine, dosing 825 mg twice daily) and PRRT to a cumulative renal AD (absorbed dose) limit of 30 Gy and dosimetry-based PRRT.
  .
  Interventions: Drug: 177Lu-DOTATOC; Drug: Capecitabine
- 177Lu-DOTATOC (Experimental): Intravenous infusion for about 7 treatment cycles with 7.5 GBq 177Lu-DOTATOC with an interval of 10 ± 2 weeks and PRRT to a cumulative renal AD limit of 30 Gy and dosimetry-based PRRT.
  Interventions: Drug: 177Lu-DOTATOC
- Standard 177Lu-DOTATOC (Active Comparator): Standard treatment of 177Lu-DOTATOC with treatment for 4 cycles.
  Interventions: Drug: 177Lu-DOTATOC

INTERVENTIONS:
Drug: 177Lu-DOTATOC — The investigational medicinal product (IMP) is 177Lu-DOTATOC which is registered as an orphan drug by the EMA ( European Medicines Agency) for the treatment of GEP-NEN (gastro-entero-pancreatic neuroendocrine tumor).
  The IMP will be administered to participants both in the control arm and the experimental arms, but with different intervals, but the same activity; 7.5 Gbq per dosing.
Drug: Capecitabine — Will be given orally with a dose of 825/m2 twice daily, starting on day 1 of each of the 4 first treatment cycles, cycle length 3 weeks.
  Arms: 177Lu-DOTATOC + Capecitabine

SUMMARY:
There are several ways of personalizing PRRT (peptide receptor radionuclide treatment) in NEN (neuroendocrine neoplasia). Nevertheless, the current treatment regimen is not personalized. This trial aims to compare personalized PRRT to non-personalized PRRT in terms of safety, efficacy and resource demands in order to optimize treatment outcomes in an evidence-based manner in future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Presence of histologically confirmed, advanced, well-differentiated, inoperable neuroendocrine tumors (NET) of any primary tumor origin and any grade, except for pheochromocytoma and paraganglioma.
* Somatostatine receptor (SSTR)-expression in tumor lesions > basal liver uptake on 68Ga-DOTA-PET
* Radiologically progressive disease within the last 1-24 months according to common clinical criteria and confirmed by the institutional multidisciplinary conference for the treatment of NETs. The CT/MRI that shows tumor progression compared to screening/baseline must have been performed 1-24 months earlier.
* All previous anti-tumor treatment except SSA must be terminated at least 4 weeks before start of treatment within the trial.
* Measurable disease according to RECIST v 1.1
* Given the available, approved anti-tumor treatments and the specific characteristics of the patient and the tumor, the investigator judges peptide receptor radionuclide therapy (PRRT) to be the treatment of choice
* GFR > 50 ml/min/1.73 m2 as determined by iohexol- or 51Cr-EDTA clearance, calculated according to a combination of LMR18 and CAPA formulas, or equally accurate method
* Hemoglobin > 90 g/L, platelets >100 x109/L, leukocytes > 3.0x109/L, neutrophils > 1.5 x109/L, aspartate transaminase (ASAT)/alanine aminotransferase (ALAT) < 3 x ULN, bilirubin < 2 x upper limit of normal (ULN), albumin > 25 g/L
* For women of child-bearing potential, highly effective contraception should be used from the time of inclusion up to at least six months after the end of treatment (EOT) visit.

Exclusion Criteria:

* Pregnancy or lactation
* Previous treatment with PRRT
* Concomitant systemic anti-tumor therapy other than somatostatin analogue (SSA)
* Contraindications for treatment with capecitabine according to the approved label.
* Discordance between CT/MRI/18F-FDG-PET and 68Ga-DOTA-PET, with evidence of tumor lesions without uptake on 68Ga-DOTATOC.
* Any other serious, uncontrolled medical or psychiatric condition that, in the opinion of the investigator, precludes the patient from participation in the trial
* Unwillingness, or inability, to participate in any part of the trial procedures or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Median progression free survival (PFS) defined as time from randomization to radiological progression. | Before start of treatment (within 4 weeks), then every 10 +/- 2 weeks weeks, at follow up (every 3-6 month (investigators choice) until progression.
  Time to progression is evaluated by CT (computed tomography) or MRI (magnetic resonance imaging) after every 16-22 weeks.
Median progression free survival (PFS) defined as time from randomization to radiological progression. | Before start of treatment (within 4 weeks), then every 10 +/- week at follow up (every 3-6 month (investigators choice) until death.
  Time to progression is evaluated by CT (computed tomography) or MRI (magnetic resonance imaging) after every 10 +/- 2 weeks.
Median progression free survival (PFS) defined as time from randomization to radiological progression, | Before start of treatment (within 4 weeks), then every 10 +/- 2 weeks, at follow up (every 3-6 month (investigators choice) or patients withdrawal of concent.. No end can be given.
  Time to progression is evaluated by CT (computed tomography) or MRI (magnetic resonance imaging) after every 16-22 weeks.

SECONDARY OUTCOMES:
Rate of treatment-related adverse reactions | At every treatment cycle, cycle length is 10 +/-2 weeks, at treatment follow up every 3-6 month (investigators choice) until progression. No time point can be given.
  Treatment-related adverse reactions graded according to CTCAE v.5.0.
Median overall survival (OS). | From date of randomization until the date of death. Timepoint unknown, as date of death can´t be predicted.
  Median OS defined as time from randomization to death of any cause.
Progression free survival. | From time of randomization until the date of first documented progression. Is evaluated within 4 weeks before randomization, after each treatment, every 10 +/2 weeks. Timepoint unknown, as date of progression can´t be predicted.
  Median progression free survival (PFS).
Percent change in sum of longest diameters (SLD) of tumor lesions. | At each radiological investigation with CT or MRI of thorax and abdomen. Is done every 10 +/- 2 weeks. In the follow up period, evaluations are done every 3-6 months until death.
  Percent change in SLD from baseline (within 4 weeks before treatment) to time of best response.
Quality of Life as judged by the patient. | Patients complete the QoL forms before start of treatment, at cycle 2 (cycle length 10+/-2 weeks), at each treatment cycle (4-approximately 7), until progression.
  All patients complete the Eastern Cooperative Oncology Group (EORTC) QoL (quality of life)-questionnaires GI- neuroendocrine tumors (NET)21.
Cumulative median absorbed dose (AD) | After each dosimetry measurements after each treatment cycle (cycle length 10 +/2 weeks), up to 18 +/-2 months.
  AD to target tumor lesions in subjects with complete remission (CR), partial remission (PR), stable disease (SD) and progressive disease (PD) as best response, according to RECIST evaluations.
Correlation between cumulative median absorbed dose and time to progression. | Every 10 +/- 2 weeks up to 18 +/- 2 months.
  Correlation between cumulative median absorbed dose to target tumor lesions and time to progression, defined as time from randomization to radiological progression.
Cumulative median absorbed dose (AD) and biological effective dose to kidneys. | Is evaluated with dosimetry after each treatment, 10 +/- 2 weeks, up to 18 +/- 2 months.
  Cumulative median AD and biological effective dose (BED) to kidneys vs rate of grade 3-4 renal toxicity (estimated and measured GFR ( glomerular filtration rate).
Differences in resource utilization and treatment cost. | Through study completion, an average of 18 months, assessed every 10 +/- 2 weeks by questionnaires.
  Differences in resource utilization and treatment cost between the two treatment arms, in relation to the progressive free survival (PFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Dept. of Oncology, Gothenburg
  - Skåne University Hospital, Dept. of Oncology, Lund
  - Karolinska University Hospital, Dept. of Oncology, Stockholm
  - Accademical Hospital, Uppsala, Dept. of Oncology, Uppsala

IPD SHARING:
Plan to Share IPD: No